CLINICAL TRIAL: NCT00456534
Title: The Effect of Smoking on Perception
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American University (Other)
Other Study IDs: Study 014
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Nicotine Dependence
Keywords: Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the experiment is to examine the effect of smoking on how individuals recognize and interpret sensory information.

DETAILED DESCRIPTION:
Participation requires one 90-minute visit on the American University campus that involves completing questionnaires and computer tasks, watching a film, and smoking a cigarette. Participants earn 30 dollars.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18 and 60
* Regular, daily smoker
* Smoke for at least 1 year

Exclusion Criteria:

* Color Blind
* Smoking Related Health Problems (Chronic Bronchitis, Chronic Obstructive Pulmonary Disease, Emphysema)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130
Dates: Start 2006-11; Study Completion 2007-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fucito, M.A., Principal Investigator — American University
Locations (1):
- American University, Dept. of Psychology, Washington D.C., District of Columbia, United States